CLINICAL TRIAL: NCT05741723
Title: OCS DCD Heart + CAP Continued Follow-Up Post-Approval Study
Brief Title: OCS DCD Heart + CAP Continued Follow-Up
Status: Active, not recruiting | Type: Observational
Sponsor: TransMedics (Industry)
Responsible Party: Sponsor
Other Study IDs: OCS-HEART-03-PAS
Record Dates: First submitted 2023-02-13; First posted 2023-02-23 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Heart Transplant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: OCS Heart — Transplanted with OCS preserved heart.

SUMMARY:
The objective of this post-approval study is to evaluate long-term outcomes of patients enrolled in the OCS DCD Heart and OCS DCD Heart CAP studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients transplanted in the OCS DCD Heart Trial and OCS DCD Heart CAP trials.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients transplanted in the OCS DCD Heart Trial and OCS DCD Heart CAP will comprise the patient population for this PAS.
Sampling Method: Non-Probability Sample
Enrollment: 276 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Patient survival | 5 years post-transplant
  Patient survival through 5 years post-transplant

OTHER OUTCOMES:
Cardiac related patient survival | 5 years post-transplant
  Cardiac related patient survival through 5 years post-transplant
Graft survival | 5 years post-transplant
  Graft survival through 5 years post-transplant
Patient and graft survival | 5 years post-transplant
  Patient and graft survival through 5 years post-transplant

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - University of California San Diago, La Jolla, California
  - Stanford University, Palo Alto, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Mayo Clinic Florida, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Northwestern Medicine, Chicago, Illinois
  - St. Vincent Cardiovascular Research Institute, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Nyph/Cumc, New York, New York
  - Montefiore, The Bronx, New York
  - Duke University, Durham, North Carolina
  - Vanderbilt Medical Center, Nashville, Tennessee
  - Sentara, Norfolk, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin